CLINICAL TRIAL: NCT04208711
Title: Study of the Role of PLA2G1B in the Immunopathogenicity by Action on CD4 T Cells During HIV Infection
Brief Title: Role of PLA2G1B During HIV Infection
Acronym: PREDIACC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diaccurate SAS (Industry)
Collaborators: CIC 1417 Cochin-Pasteur (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PREDIACC; 2018-A02025-50 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2019-12-02; First posted 2019-12-23 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: HIV Infections
Keywords: HIV infection; PLA2G1B; Lymphocyte CD4+
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- positive HIV patient not treated by ARV yet (Other): Before starting HIV treatment, 15 patients will be included in the study and 50mL of whole blood will be taken. After treatment initiation 8 of the 15 patients will entered in the follow-up phase for 1 year (5 followup visit, M1, M3, M6, M9, M12) and 30mL of whole blood will be taken at each visit.
  The duration of the study for the 7 other patients will be 1 day.
  Interventions: Other: biological sample

INTERVENTIONS:
Other: biological sample — whole blood sample

SUMMARY:
The main objective of this study is to qualify and quantify, by microscopy techniques, CD4+ lymphocyte abnormalities during HIV infection in 7 patients who are naive to any ARV (antiretroviral ) treatment and secondarily to follow the kinetics of reversion of the observed abnormalities, as well as the evolution of the levels of PLA2G1B and its cofactor gp41 in 8 patients under ARV treatment

DETAILED DESCRIPTION:
Antiretroviral therapy in HIV-infected patients has progressed significantly over the past two decades.

Viral replication in patients who are complicit in their treatment regimen is greatly reduced below detection limits (quantification) by current and approved laboratory tests. However, the persistence of residual (plasma) replication of the virus creates an inflammatory state associated with certain pathologies, accelerated aging and premature mortality. If treatment is discontinued for any reason, viral replication resumes within a few weeks in almost all patients.

Alternative infections of inflammatory pathways in HIV can also play a critical role in the inflammatory process suppressed by treatment. Members of the phospholipase A2 family can hydrolyze phospholipid molecules at the sn-2 position, making it a question about lipid moieties. One of the members, the phospholipase A2 group1B (PLA2G1B), is found in the plasma of HIV-infected patients who are not receiving antiretroviral therapy. Ex vivo, this enzyme is able to induce a purified CD4 lymphocyte energy from donors, as well as by inducing the lack of response to IL-7 (interleukin-7). In the long term, loss of response to IL-7 induces CD4 lymphopenia. Therefore, PLA2G1B must play an important role in the mechanism leading to HIV-infected patients becoming immunodeficient.

At the clinical level, we found that PLA2G1B activity increases in all HIV-infected patients and decreases after ARV treatment. On the other hand, for patients who are able to eliminate the HIV virus on therapy but whose immunological response remains low, PLA2G1B activity remains high. More interestingly, in "HIV Elite Controller" patients, PLA2G1B activity is not found in their plasma. Overall, there is a correlation between the different clinical groups (viremic not on therapy, ARV and virus removal with robust CD4+ T-cell response, virus removal with suboptimal CD4+ T-cell response and "HIV Elite Controller") and the activity level of PLA2G1B in their plasma.

The purpose of this study, more generally, is to study the role of PLA2G1B in CD4 lymphocytes and to analyze the reversion of its effects in the immunopathogenicity of HIV infection.

In the main study, 15 patients will be included. The analysis of the first 7 patients will in addition meet the objectives of the study, to determine the test that will allow the follow-up of the 8 other patients after ARV treatment. The participation of the 7 patients in the study is limited to 1 (one) day.

In the sub-study, the last 8 patients following their inclusion in the main study will enter a follow-up phase of 12 months after they are put on ARV treatment. The total duration of participation for the 8 patients will be 13 months.

The main study is carried out by taking 50 mL of total blood and in the sub-study, 30mL of blood sample will be taken during the follow-up visit (at M1, M3, M6, M9 and 12 Months) after ARV treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participant aged 18 to under 70
2. Participant having signed the written and informed consent;
3. Patient with HIV-1 infection documented by a positive HIV western blot positive (infected patients> 6 months, CD4 count> 350 / mm3 and HIV RNA <100.000 copies / mL) naive to any ARV treatment Anti-HIV antibody positive and an optical density <1.0, as determined by enzyme immunoassay, with no significant risk of clinical events
4. Appropriate laboratory data: hemoglobin> 9 g / dL, absolute neutrophil count ≥1000 / μL, platelets ≥50,000 / μL, bilirubin ≤ 1.5 X upper limit of normal (ULN) or ≤3 X ULN serum creatinine ≤ 1.5 X ULN, alanine amino transferase (ALT) or aspartate amino transferase (AST) ≤ 3 X ULN;
5. ECOG (Eastern Cooperative Oncology Group) performance status scale ≤2
6. Subject benefiting from a French social security scheme, or affiliated to such a scheme

Exclusion Criteria:

1. History of inflammatory disease such as rheumatoid arthritis, lupus, Crohn's disease, ulcerative colitis
2. Concomitant use of systemic or topical corticosteroids for the treatment of skin diseases. However, topical steroids and oral steroids (≤10 mg prednisone equivalent / day) are permitted if the patient has received a stable dose with stable symptoms for at least 4 weeks before inclusion in the study.
3. Major surgery <4 weeks before inclusion in the study.
4. A stem cell transplant.
5. History of other malignancies in the last three years except Kaposi controlled.
6. Infection known by hepatitis C or B virus (HCV or HBV)
7. Congestive heart failure, class III or IV, according to the criteria of the New York Heart Association (NYHA).
8. Vulnerable population (minors, pregnant, parturient or nursing women, persons under guardianship or trusteeship, or deprived of liberty by a judicial or administrative decision, under the protection of justice)
9. Patients with dementia or altered mental states who would not understand and provide an informed consent document

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
immunological : to qualify and quantify by confocal microscopic techniques and flow cytometry lymphocyte abnormalities | up to 1 year
  The assessment of the change in the proportion of lymphocytes at 1, 3, 6, 9 and 12 months as compared to Day 1:
  * CD4 with membranes abnormalities above normal,
  * CD4 with major membrane abnormalities,
  * CD4 with signal transduction abnormalities,
  * CD4 reversing one of these abnormalities spontaneously or after treatment with neutralizing monoclonal antibody (mAb) 2B2

SECONDARY OUTCOMES:
immunological | up to 1 year
  The assessment by immunophenotyping test ( flow cytometry) of the change at 1, 3, 6, 9 and 12 months as compared to Day 1 of:
  * number of CD4/mm3 of blood, number of CD8/mm3 of blood, CD4 / CD8 ratio, viral load (copies of HIV RNA/mL of blood), viral DNA (copies of HIV DNA/mL of blood)
  * number of CD4/mm3 secreting IFN gamma (Interferon gamma), TNF (Tumor necrosis factor) and IL-2 (Interleukin-2) (in % of IFN - TNFa - IL-2+ / CD4)

CONTACTS AND LOCATIONS:
Overall Officials: Odile LAUNAY, MD, PHD, Principal Investigator — CIC 1417 Clinical Center Investigation - Cochin Hospital, AP-HP
Locations (1):
- CIC 1417 Cochin Pasteur, hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No